CLINICAL TRIAL: NCT05900388
Title: Xarelto Paediatric VTE PASS Drug Utilization Study: An Observational, Longitudinal, Multi-source Drug Utilization Safety Study to Evaluate the Drug Use Patterns and Safety of Rivaroxaban Oral Suspension in Children Under Two Years With Venous Thromboembolism
Brief Title: A Study to Observe the Pattern of Use and Safety of Rivaroxaban in Children Under 2 Years Old With Venous Thromboembolism (VTE)
Acronym: XAPAEDUS
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 22195
Record Dates: First submitted 2023-05-10; First posted 2023-06-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism; Children Under 2 Years
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with VTE: Pediatric patients under two years who initiate an anticoagulation therapy with rivaroxaban oral suspension or Standard of care (SOC) following a VTE diagnosis.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Standard of care (SOC)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Retrospective cohort analysis using National health registers in Denmark and Sweden; Système National Des Données De Santé (SNDS) in France and Sistema d'Informació per al Desenvolupament de l'Investigació en Atenció Primària (SIDIAP) in Spain
Drug: Standard of care (SOC) — Retrospective cohort analysis using National health registers in Denmark and Sweden; Système National Des Données De Santé (SNDS) in France and Sistema d'Informació per al Desenvolupament de l'Investigació en Atenció Primària (SIDIAP) in Spain. SOC including heparins, Vitamin K antagonists (VKAs) and Other Direct oral anticoagulants (DOACs).

SUMMARY:
This is an observational study in which only data are collected from participants receiving their usual treatment. The study is done in children under 2 years old with venous thromboembolism (VTE).

VTE is a condition in which blood clots form in the veins, usually in the leg. This can cause pain and swelling. The clot can also break apart and travel in the blood to the lungs where it can block the blood flow. This can be life threatening.

Rivaroxaban is approved for doctors to prescribe to children with VTE, but there is limited information about how it is used, how well it works, and how safe it is in children under 2 years old. Children in this study are already receiving or will receive rivaroxaban or other currently used medicines for VTE from their doctor according to the approved product information.

The purpose of this study is to collect information on the pattern of use and safety of rivaroxaban and other standard medicines for VTE in children under 2 years old.

The main information that researchers will collect in this study:

* Age, gender, and other information about the child and their illness
* Type of VTE treatment given to the child
* Occurrence of medically important bleeding and its severity

Further information that researchers will collect:

* Changes in the characteristics of the children given VTE treatment (e.g., changes in the age range of children given VTE treatment) and changes in the treatment pattern for VTE
* Return of VTE symptoms
* Types of doctors who prescribe VTE treatment and their set-up (e.g., special clinics versus hospitals) Besides this data collection, no further tests or examinations are needed in this study.

The data for this study will be collected from electronic health records and health insurance claims data until 2026.

Researchers will observe each child during treatment until:

* end of the anticoagulation treatment period e.g. discontinuation of all study drugs,
* their information is no longer available, or
* the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of initiation of an anticoagulant therapy (index drug), either rivaroxaban oral suspension or other anticoagulation therapies (heparins, Vitamin K antagonists (VKAs), other Direct oral anticoagulants (DOACs)). Initiation will be defined as a first record of any anticoagulation therapy (rivaroxaban or SOC) without any anticoagulation therapy in the previous 6 months, or since date of birth for children less than 6 months
* Evidence of a prior VTE diagnosis (index VTE), defined as the presence of at least one primary/main or secondary diagnosis code for VTE recorded in inpatient setting in the previous 30 days
* Age less than two years on index date.
* Baseline period for availability of patient data history in the data source. A minimal baseline period of six months before index date for children aged between six months and two years, and a baseline period since birth for children less than six months of age will be required.

Exclusion Criteria:

- None

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged under two years who initiate an anticoagulation therapy with rivaroxaban oral suspension or any other anticoagulation drug (index date) following a VTE diagnosis during year 2021 to 2026.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive summary of demographic characteristics of patients | Retrospective data analysis from 2021 to 2026
Descriptive summary of characteristics of index venous thromboembolism (VTE) | Retrospective data analysis from 2021 to 2026
Co-morbidities reported in the previous six months before index date, or since date of birth for children less than six months | Retrospective data analysis from 2021 to 2026
Prior treatments reported in the previous six months before index date (or since date of birth for children less than six months) | Retrospective data analysis from 2021 to 2026
Comedication during follow-up | Retrospective data analysis from 2021 to 2027
Descriptive summary of Health resource utilization in the previous six months before index date (or since date of birth for children less than six months) | Retrospective data analysis from 2021 to 2026
Duration of oral, nasogastric/gastric feeding before index date, if available | Retrospective data analysis from 2021 to 2026
Substance and class of anticoagulant drug therapy | Retrospective data analysis from 2021 to 2027
  For analyzing Index drug therapy and Maintenance therapy.
Duration of use anticoagulant drug therapy | Retrospective data analysis from 2021 to 2027
  For analyzing Index drug therapy and Maintenance therapy.
Dosing of anticoagulant drug administration | Retrospective data analysis from 2021 to 2027
  For analyzing Index drug therapy and Maintenance therapy.
Route of anticoagulant drug administration | Retrospective data analysis from 2021 to 2027
  For analyzing Index drug therapy and Maintenance therapy.
Switching to other anticoagulant therapy (Yes/No) | Retrospective data analysis from 2021 to 2027
Number of successive anticoagulation agents during an anticoagulant treatment period | Retrospective data analysis from 2021 to 2027
Sequence of successive anticoagulation agents during an anticoagulant treatment period | Retrospective data analysis from 2021 to 2027
Incidence and severity of major bleeding according to anticoagulation therapy | Retrospective data analysis from 2021 to 2027
Incidence and severity of clinically Relevant Non-Major (CRNM) bleeding according to anticoagulation therapy | Retrospective data analysis from 2021 to 2027

SECONDARY OUTCOMES:
Time trends by calendar year in patient characteristics | Retrospective data analysis from 2021 to 2026
  Description by calendar year of age group at index date and medical history at index date.
Time trends by calendar year in anticoagulation treatment patterns | Retrospective data analysis from 2021 to 2026
  Description by calendar year of class of anticoagulation therapy at initiation.
Incidence of recurrent symptomatic VTE according to anticoagulation therapy | Retrospective data analysis from 2021 to 2027
Physician specialty and care settings (inpatient care, secondary outpatient care, primary care) for prescriptions of anticoagulation therapy | Retrospective data analysis from 2021 to 2027

CONTACTS AND LOCATIONS:
Locations (4):
- Many locations, Multiple Locations, Denmark
- Many locations, Multiple Locations, France
- Many locations, Multiple Locations, Spain
- Many locations, Multiple Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.